CLINICAL TRIAL: NCT01624441
Title: A Phase 1 Study With Dose Expansion of Dinaciclib (SCH 727965) in Combination With Epirubicin in Patients With Metastatic Triple Negative Breast Cancer
Brief Title: Dinaciclib and Epirubicin Hydrochloride in Treating Patients With Metastatic Triple-Negative Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-00950; NCI-2012-00950 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2012-0229 (Other: M D Anderson Cancer Center); 9138 (Other: CTEP); P30CA016672 (NIH); R01CA152228 (NIH); U01CA062461 (NIH)
Record Dates: First submitted 2012-06-18; First posted 2012-06-20 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Estrogen Receptor Negative; HER2/Neu Negative; Male Breast Carcinoma; Progesterone Receptor Negative; Recurrent Breast Carcinoma; Stage IV Breast Cancer AJCC v6 and v7; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — dinaciclib; Epirubicin

ARMS (1):
- Treatment (dinaciclib and epirubicin hydrochloride) (Experimental): Patients receive dinaciclib IV over 2 hours on day 1 and epirubicin hydrochloride IV over 30 minutes on day 2. Treatment repeats every 21 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dinaciclib; Drug: Epirubicin Hydrochloride; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Dinaciclib — Given IV
  Other Names: CDK Inhibitor SCH 727965; MK-7965; SCH 727965
Drug: Epirubicin Hydrochloride — Given IV
  Other Names: Ellence; IMI-28; Pharmorubicin PFS
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I clinical trial studies the side effects and the best dose of dinaciclib when given together with epirubicin hydrochloride (epirubicin) in patients with metastatic (cancer that has spread to other parts of the body) triple-negative breast cancer. Dinaciclib is designed to stop cancer cells from dividing into new cancer cells. Epirubicin is designed to block the way cancer cells grow and divide and may slow or stop cancer cells from spreading throughout the body. Researchers want to find out what is the highest tolerable dose of the experimental drug dinaciclib that can be given in combination with epirubicin in patients with metastatic triple negative breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of dinaciclib given in combination with epirubicin in patients with metastatic triple negative breast cancer.

SECONDARY OBJECTIVES:

I. To determine the predictive value of myeloid cell leukemia sequence 1 protein (MCL-1), low molecular weight cyclin E (LMW-E), and tumor grade as predictors of biologic response (i.e. induction of apoptosis) in tumors treated with therapy.

II. To evaluate the efficacy of combination therapy. III. To determine the effects of therapy on proliferation as measured by proliferation-related Ki-67 antigen (Ki67) and apoptosis as measured by terminal deoxynucleotidyl transferase (TdT)-mediated dUTP nick end labeling assay (TUNEL).

OUTLINE: This is a dose-escalation study of dinaciclib.

Patients receive dinaciclib intravenously (IV) over 2 hours on day 1 and epirubicin hydrochloride IV over 30 minutes on day 2. Treatment repeats every 21 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed estrogen receptor (ER)/progesterone receptor (PR)/human epidermal growth factor receptor 2 (HER2) negative carcinoma of the breast that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective; for purposes of this study, triple negative disease will be tumors that have ER/PR < 10% and HER2 =< 1+ by immunohistochemistry (IHC) or HER2 fluorescent in situ hybridization (FISH) non-amplified (ratio < 2)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Patients must have no more than two prior chemotherapy regimens for metastatic breast cancer; in patients who develop disease recurrence within 6 months of adjuvant or neoadjuvant chemotherapy, the adjuvant or neoadjuvant therapy will be considered one prior regimen for metastatic disease
* Life expectancy of greater than 3 months
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal limits unless clinical diagnosis of Gilbert's syndrome
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Patients must be disease free of prior malignancy for >= 5 years with the exception of curatively treated squamous cell carcinomas of the skin or carcinoma in situ of the cervix or breast
* Must have at least one site of objective measurable or evaluable disease; baseline measurements and evaluations must be obtained within 4 weeks of start of therapy
* Patients must have no history of prior therapy with dinaciclib
* Concurrent use of hormonal therapy is not permitted; concurrent radiation therapy is not permitted; bisphosphonates are allowed, provided that they were started no less than two weeks prior to initiating protocol therapy
* Patients must have completed and recovered from the effects of prior chemotherapy (< grade 2 toxicity) excluding alopecia
* Women of child-bearing potential and men must agree to use adequate contraception (barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of dinaciclib administration
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events
* Patients who are receiving any other investigational agents
* Patients with untreated brain metastases should be excluded from this clinical trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition as epirubicin or dinaciclib
* Patients receiving any medications or substances that are inhibitors or inducers of cytochrome P450 family 3, subfamily A, polypeptide 4/5 (CYP3A4/5) are ineligible
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with dinaciclib
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Patients who have had prior organ allograft or require immunosuppressive therapy
* Patients who have received a cumulative dose of doxorubicin of greater than 360 mg/m^2 or epirubicin of greater than 600 mg/m^2; patients who have received > 240 mg/m^2 of doxorubicin or > 400 mg/m^2 of epirubicin should be advised to undergo evaluation of left ventricular ejection fraction (LVEF) with echocardiogram or multi gated acquisition scan (MUGA) prior to initiating therapy
* Patients with a history of New York Heart Association class 3 or 4 heart failure, or history of myocardial infarction, unstable angina or cerebral vascular accident (CVA) within 6 months of protocol registration
* LVEF < 50% by MUGA or echocardiogram (ECHO)
* Patients who have history of PR prolongation or atrioventricular (AV) block

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-08-21 (Actual); Primary Completion 2013-09-10 (Actual); Study Completion 2013-09-10 (Actual)

PRIMARY OUTCOMES:
MTD of dinaciclib given in combination with epirubicin hydrochloride, determined according to incidence of dose-limiting toxicity (DLT) graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4 | 21 days
  The number (%) of DLTs will tabulate by dose level of dinaciclib.

SECONDARY OUTCOMES:
Predictive value of MCL-1, LMW-E, and tumor grade as predictors of biologic response (i.e. induction of apoptosis) in tumors treated with therapy | Up to 30 days after completion of study treatment
  A logistic regression model will be used to assess whether the expression level of LMW-E can predict clinical benefit, adjusted for dose level and other potential prognostic factors: visceral organ involvement (present vs. absent), number of prior therapies for metastatic breast cancer (0-2 or > 2), age (< 60 vs. > 60) and ECOG performance status (0-1 vs. 2).
Clinical benefit rate (complete response [CR] + partial response [PR] + stable disease [SD]), assessed using Response Evaluation Criteria in Solid Tumors (RECIST) | At 6 months
  The overall clinical benefit rate for patients treated at the MTD will be estimated with a 90% credible interval.
Changes in proliferation as measured by Ki67 and apoptosis as measured by TUNEL | From baseline to 2 weeks
  For the patients with pre- and post- treatment biopsies, summary statistics used to describe change in apoptotic index pre- to post-treatment, and boxplots to illustrate distribution pre- and post-treatment, as well as distribution of change. Mean change estimated with 95% confidence interval. MCL-1, LMW-E, and Ki67 similarly analyzed. Analyses also performed stratified by tumor grade. Correlation between changes in MCL-1 and LMW-E pre- to post-treatment estimated with 95% confidence interval. Number of tumors in 4 categories (negative, low, medium, high) tabulated by % of TUNEL+ tumor cells.

CONTACTS AND LOCATIONS:
Overall Officials: Stacy Moulder, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Mitri Z, Karakas C, Wei C, Briones B, Simmons H, Ibrahim N, Alvarez R, Murray JL, Keyomarsi K, Moulder S. A phase 1 study with dose expansion of the CDK inhibitor dinaciclib (SCH 727965) in combination with epirubicin in patients with metastatic triple negative breast cancer. Invest New Drugs. 2015 Aug;33(4):890-4. doi: 10.1007/s10637-015-0244-4. Epub 2015 May 7. PMID 25947565